CLINICAL TRIAL: NCT03453203
Title: Treatment of Cervical Pain in Chronic Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHClevelandMC1
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Chronic Migraine
Keywords: Chronic migraine; Osteopathic manipulative treatment; Cervicalgia
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Blinded control trial
Who Masked: Care Provider
Masking Description: The follow-up physician will be blinded to treatment vs control arm. Patient will be selected randomly depending on the time of recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Both arms with be diagnosed using tenderpoints In the control arm the tenderpoint will Be palpated for 90 secs with no counterstrain treatment applied.
  Both treatment and control groups will remain on their current migraine medication regiment.
  Interventions: Other: Osteopathic Manipulative Treatment Using Counterstrain
- Treatment (conterstrain) (Other): Both arms with be diagnosed using tenderpoints. Treatment arm will be treated with counterstrain technique. Counterstrain is a passive manipulative technique which the tissue being treated is positioned at a point of balance, or ease, AWAY from the restrictive barrier (The most thought of form of manipulative technique is high velocity low amplitude which is typically performed by chiropractors in spinal manipulation which goes TOWARD the restrictive barrier and actually pass through the restrictive barrier). Once a tenderpoint is found in the muscles the area of treatment is placed in a (three dimensional) position that will eliminate the sensation (tenderness).The treatment position is held for 90 seconds or until a release is felt (a decrease in muscle tension). Both treatment and control groups will remain on their current migraine medication regiment.
  Interventions: Other: Osteopathic Manipulative Treatment Using Counterstrain

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment Using Counterstrain — Described in arm/group descriptions
  Other Names: Strain/Counterstrain

SUMMARY:
Chronic migraine (CM) is defined as a headache that occurs more than 15 days per month, which has the features of migraine headache on at least 8 days per month.1 The cause of CM is not well understood. Many patients with CM appear to have associated musculoskeletal neck pain. The purpose of this study is to treat cervicalgia in patients with migraine and to look for improvement in migraine frequency and intensity. Osteopathic manipulative treatment (OMT) can diagnose and treat common musculoskeletal dysfunction. This may break facilitation within the nervous system and reduce musculoskeletal pain which subsequently will reduce headache frequency. This will be a randomized controlled trail comparing patients with CM treated with OMT vs no treatment. The investigators will look at the frequency of migraine days before and after the treatment period to determine migraine frequency and improvement.

DETAILED DESCRIPTION:
Data will be analyzed by reviewing the amount of headache days during the treatment period

Patients will be distributed randomly into either the treatment arm or control arm. Subjects will be randomized as they are recruited for the study (i.e. subject 1 treatment, subject 2 control, subject 3 treatment, etc.) The participants will be distributed by a research assistant who will allocate the patients randomly to one of the two arms.

Both arms will be diagnosed using tenderpoints (Tenderpoints are small tense edematous areas of tenderness about the size of a fingertip. They are typically located near bony attachments of tendons, ligaments, or in the belly of some muscles).Tenderpoints will be documented and stored in a secure flash drive.

Treatment arm will be treated with an Osteopathic manipulative treatment called counterstrain technique. Osteopathic manipulative treatment is a hands on palpation of the tissues to diagnose and treat neuromusculoskeletal dysfunction. Counterstrain is a passive manipulative technique which the tissue being treated is positioned at a point of balance, or ease, AWAY from the restrictive barrier (The most thought of form of manipulative technique is high velocity low amplitude which is typically performed by chiropractors in spinal manipulation which goes TOWARD the restrictive barrier and actually pass through the restrictive barrier). Once a tenderpoint is found in the muscles the area of treatment is placed in a (three dimensional) position that will eliminate the sensation (tenderness).The treatment position is held for 90 seconds or until a release is felt (release is usually a decrease in the tone or muscle tension).

In the control arm the tenderpoint will Be palpated for 90 seconds with no counterstrain treatment applied. (Risk are possible soreness at palpation site though not likely, there is no benefit) Both treatment and control groups will remain on their current migraine medication regiment.

They will follow-up with Dr. Deborah Reed, MD, FAHS who is a board certified neurologist and headache specialist. This investigator will be blinded to weather the patient received counterstrain manipulation or no treatment. The investigator will document the number of headache days between follow-up periods.

After the first treatment follow-up will occur as follows: Week 1, Week 2, Week 4, Week 6, Week 10. This is picked somewhat arbitrarily as typical treatment follow-ups will vary from patient to patient depending on the severity of the musculoskeletal dysfunction (somatic dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years of age who fit the ICHD-3 criteria for Chronic Migraine. These patients must be currently on an abortive agent (such as a triptans, NSAIDs) and require at least 8 doses a month.

Exclusion Criteria:

* Patients will be excluded if there are any signs of secondary headaches. If they have received BOTOX therapy in the past 4 months or are currently receiving BOTOX therapy. If the patients have contraindications to counterstrain OMT (clinical signs of Fractures, ligament instability, severe vertebral artery disease) or are a poor candidate for OMT (unable to follow commands, unable to fully relax).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-29 (Estimated); Primary Completion 2018-12-29 (Estimated); Study Completion 2018-12-29 (Estimated)

PRIMARY OUTCOMES:
Treatment of Cervical Pain in Chronic Migraine | 3 months
  Frequency of migraine days after treatment with Osteopathic manipulative treatment using counterstrain